CLINICAL TRIAL: NCT03988946
Title: Cephea Mitral Valve and Transseptal Delivery System FIH
Brief Title: Cephea Transseptal Mitral Valve System FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cephea Valve Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP21549
Record Dates: First submitted 2019-01-10; First posted 2019-06-18 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Transcatheter Mitral Valve Replacement (Experimental): Replacement valve delivered through a transfemoral access and transseptal approach
  Interventions: Device: Transcatheter Mitral Valve Replacement via Transseptal Access

INTERVENTIONS:
Device: Transcatheter Mitral Valve Replacement via Transseptal Access — The Cephea Transseptal Mitral Valve System is intended for use in symptomatic patients with moderate to severe degenerative or functional mitral regurgitation, who are poor candidates for surgery and who are anatomically eligible for the treatment.

SUMMARY:
To assess the safety and performance of the Cephea Transseptal Mitral Valve System for the treatment of symptomatic moderate to severe degenerative or functional mitral regurgitation, in patients who are poor candidates for surgery.

ELIGIBILITY:
MVARC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Safety as measured by freedom from major adverse events | 30 days
  Freedom from major adverse events, including:
  * All-cause mortality
  * Disabling stroke
  * Myocardial infarction
  * Renal failure requiring dialysis
  * Life-threatening bleeding
  * Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention.
Performance | 30 days
  Reduction in mitral regurgitation to ≤1+

CONTACTS AND LOCATIONS:
Overall Officials: Helen J Scotch, Study Director — Cephea Valve Technologies
Locations (1):
- St. Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided